CLINICAL TRIAL: NCT05312281
Title: Prospective Randomised Study Comparing Postoperative Treatment After Surgical Decompression for Lumbar Spinal Stenosis. With and Without Immobilisation in an Orthosis
Brief Title: Study Comparing Postoperative Treatment After Surgical Decompression for Lumbar Spinal Stenosis.
Acronym: SURGIMMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SRH Gesundheitszentrum Bad Herrenalb (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GBH-O1
Record Dates: First submitted 2022-03-10; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group "without lumbar belt" (No Intervention): Control group "without lumbar belt"
- Device : Lombastab immo. wear for 6 weeks post-surgery the Lombastab Immo (Experimental): Lombastab immo. wear for 6 weeks post-surgery the Lombastab Immo
  Interventions: Device: Device : Lombastab immo. wear for 6 weeks post-surgery the Lombastab Immo

INTERVENTIONS:
Device: Device : Lombastab immo. wear for 6 weeks post-surgery the Lombastab Immo — Wear for 6 weeks post-surgery
  Arms: Device : Lombastab immo. wear for 6 weeks post-surgery the Lombastab Immo

SUMMARY:
The aim of the study is to assess the benefit of wearing a lumbar orthosis after surgery for spinal stenosis. It will be evaluated if a post-surgery immobilization for 6 weeks with a lumbar orthosis reduces early recurrence, increases walking distance, decreases significantly faster pain and pain medication after surgery

DETAILED DESCRIPTION:
Spinal stenosis and orthoses The study situation in this regard is very poor, high-quality level 1 studies are not available.

A study by Prateepavanich et al. from 2001 shows advantages in the therapy with lumbar orthoses in neurogenic spinal claudication in the context of conservative therapy (9). Regarding postoperative prescription, expert opinions have long diverged (10). Nevertheless, in a survey of North American spine surgeons, over 60% reported prescribing an orthosis postoperatively (11).

2 Aim of the study

The aim of this study is to show that patients after surgical decompression for lumbar spinal stenosis and patients after surgical sequestrectomy benefit from temporary postoperative immobilization using a lumbar orthosis.

To show that postoperative therapy with a lumbar orthosis prolongs walking distance and reduces early recurrence.

It will be shown that postoperative pain decreases significantly faster and thus pain medication can be reduced faster early postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Decompression with hemi-/ partial laminectomy, one. Laminectomy, and foraminotomy. Flavectomy with undercutting due to uni-and multi-segmental spinal stenosis.
* Age 20-80 years
* Pre-operative walking distance at least 100m
* Consent form signed by the patient

Exclusion Criteria:

* Fusion surgery or recurrent surgery
* Tumors of the spine
* Cervical spinal stenosis or myelopathy
* Rheumatoid arthritis or similar autoimmune disease
* Infection - request for a pension
* Dyspnea due to heart failure with limited walking distance
* Peripheral Arterial Occlusive Disease (PAOD)-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-06-28 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate or reherniation/restenosis by means of MRI results | at 104 weeks
  symptomatic reduction of Walking distance

SECONDARY OUTCOMES:
Pain and Disability Index | At 0, 2, 6, 12, 24, 52 and 104 weeks
  Visual analog scale (VAS) (visual analog scale of 0-10, 0 means no pain, 10 means extreme pain, we expect better outcome with Lombastab), Oswestry Disability Questionaire (german version scale of 0-50, 0 means no impairment at all, 50 means highest possible impairment, we expect lower impairment due to Lombastab)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Veihelmann, Prof, Study Chair — SRH Ges.-Zentrum Bad Herrenalb
Locations (1):
- Klinikum Karlsruhe, Karlsruhe, Germany